CLINICAL TRIAL: NCT05637125
Title: Effect of Different Types of Aerobic Training on Peak VO2 and Ejection Fraction for Diastolic Heart Failure Patients; a Comparative Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Tamer Ibrahim Abo Elyazed, Ass.prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BeniSuefU2
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Effect of Different Types of Aerobic Training on Diastolic Heart Failure Patients
Keywords: Diastolic heart failure; ejection fraction; aerobic exercise; peak VO2
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A received aerobic exercise for upper limb in the form of arm ergometer 3 session/week for 12 weeks.
  Interventions: Other: aerobic exercise for upper limb
- Group B (Active Comparator): received aerobic exercise for lower limb in the form of cycling 3session/week for 12 weeks.
  Interventions: Other: aerobic exercise for lower limb

INTERVENTIONS:
Other: aerobic exercise for upper limb — aerobic exercise for upper limb in the form of arm ergometer 3 session/week for 12 weeks. Patient started with warming up for 5 minutes in form of stretching. Patients used arm ergometer without resistance for upper limb aerobic exercise for 20 minutes and instructed to take rest if they feel tired or fatigue. The intensity was according to rate of perceive exertion, after 20 minutes, patients were asked to cool down for 5 minutes in the form of stretching at the end of an exercise session.
  Arms: Group A
Other: aerobic exercise for lower limb — received aerobic exercise for lower limb in the form of cycling 3session/week for 12 weeks. Patient started with warming up for 5 minutes. Patients used bicycle for lower limb aerobic exercise for 20 minutes and instructed to take rest if they feel tired or fatigue. The intensity was according to rate of perceive exertion. After 20 minutes, patients were asked to cool down for 5 minutes in the form of stretching at the end of an exercise session.
  Arms: Group B

SUMMARY:
Background: Heart failure is described by a lack of confirmed efficient therapies and exercise intolerance. Physical activity is related to a lower risk of adverse cardiovascular consequences, involving heart failure. The purpose of the study: determine the effect of different types of aerobic training on peak VO2 and ejection fraction in diastolic heart failure patients. Subject and methods: Forty eligible male patients with diastolic heart failure, aged between 50 - 60 years old, participated in this study. They were selected from an outpatient clinic of general Zagazig hospital and were assigned into 2 equal groups in numbers. The first group (A) received aerobic exercise for the upper limb in form of arm ergometer exercises, while the second group (B) received aerobic exercise for the lower limb in form of cycling. Training duration for both groups was 3 sessions/week for 12 weeks. Peak VO2, and ejection fraction of both groups were measured and compared pre and post-treatment. Results: There was no significant difference in the ejection fraction between groups post-treatment. There was a significant increase in the peak VO2 of group B compared with that of group A post-treatment. Conclusion: there is no effect of different types of aerobic training on ejection fraction and peak VO2 for diastolic heart failure patients, but lower limb exercise is more effective than upper limb exercise in improvement of peak VO2 for diastolic heart failure patients.

DETAILED DESCRIPTION:
Ejection fraction and peak VO2 of both groups were measured pre exercise program and after 12 weeks at the end of the study exercise program.

* Vivid S5 cardiovascular ultrasound system (BT308), made in china, was used to measure ejection fraction.
* Oxycon pro (ER900, Germany) cardiopulmonary exercise test unit was used to measure Peak Vo2

Treatment procedure:

Group A received aerobic exercise for upper limb in the form of arm ergometer 3 session/week for 12 weeks. Patient started with warming up for 5 minutes in form of stretching. Patients used arm ergometer without resistance for upper limb aerobic exercise for 20 minutes and instructed to take rest if they feel tired or fatigue. The intensity was according to rate of perceive exertion, after 20 minutes, patients were asked to cool down for 5 minutes in the form of stretching at the end of an exercise session.

Group B received aerobic exercise for lower limb in the form of cycling 3session/week for 12 weeks. Patient started with warming up for 5 minutes. Patients used bicycle for lower limb aerobic exercise for 20 minutes and instructed to take rest if they feel tired or fatigue. The intensity was according to rate of perceive exertion. After 20 minutes, patients were asked to cool down for 5 minutes in the form of stretching at the end of an exercise session.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* under complete medical supervision
* left ventricular end diastolic dimension >5.5cm
* ejection fraction <50%.

Exclusion Criteria:

* Orthopedic problems
* Mental disorders
* Metabolic disorders (D.M)
* Current treatment for cancer or active infection.

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | 12 weeks
  Vivid S5 cardiovascular ultrasound system (BT308), made in china, was used to measure ejection fraction.
peak VO2 | 12 weeks
  Oxycon pro (ER900, Germany) cardiopulmonary exercise test unit was used to measure Peak Vo2

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Abo Elyazed, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Banī Suwayf, Sharq, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obaya HE, El-Moneim Abd El-Hakim AA, Fares HM, Eldin Saad MK, Abo Elyazed TI. Effect of different types of aerobic training on peak VO2 and ejection fraction for diastolic heart failure patients; a comparative randomized control trial. Physiother Res Int. 2024 Jan;29(1):e2044. doi: 10.1002/pri.2044. Epub 2023 Aug 3. PMID 37537847